CLINICAL TRIAL: NCT00228410
Title: A Multicenter, Randomized, Double-Blind Comparison of the Safety and Efficacy of Tigecycline With Those of Vancomycin With Aztreonam to Treat Complicated Skin and Skin Structure Infections in Hospitalized Patients.
Brief Title: Study Comparing Tigecycline and Vancomycin With Aztreonam in Complicated Skin and Skin Structure Infections
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3074A1-305
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Skin Diseases, Infectious
Keywords: Skin Infections; Skin Disease
MeSH Terms: conditions — Skin Diseases, Infectious; Cellulitis; Skin Diseases | interventions — Tigecycline; Vancomycin; Aztreonam

INTERVENTIONS:
Drug: Tigecycline
Drug: vancomycin with aztreonam

SUMMARY:
To compare the safety and the efficacy of tigecycline to vancomycin with aztreonam in treating hospitalized patients with complicated skin and/or skin structure infections.

ELIGIBILITY:
Inclusion Criteria:

* Anticipated need for intravenous antibiotic therapy of 5 days or longer.
* Patients known or suspected to have a complicated skin and skin structure infection. Complicated skin/skin structure infection includes infections either involving deeper soft tissue or requiring significant surgical intervention or a significant underlying disease state (such as diabetes mellitus, peripheral vascular disease, peripheral neuropathy, lower venous insufficiency) that complicates response to treatment.

Other inclusion applies

Exclusion Criteria:

* Patients with any concomitant condition that, in the opinion of the investigator, would preclude an evaluation of a response or make it unlikely that the contemplated course of therapy could be completed.
* Patients with severely impaired arterial blood supply and insufficiency such that the likelihood of amputation of the infected anatomical site within one month is likely.
* Infected diabetic foot ulcers or decubitus ulcers where the infection is present for greater than one week's duration or chronically infected decubitus ulcers in patients who can not be compliant with measures necessary for chronic wound healing.
* Necrotizing fasciitis or gangrene.

Other exclusion applies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2002-11; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint was the clinical response in the co-primary populations of the clinically evaluable (CE) and clinical modified intent-to-treat (c-mITT) subjects at the test-of-cure assessment.

SECONDARY OUTCOMES:
Safety assessments included a physical examination and daily recording of vital signs (temperature, heart rate, blood pressure).

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Teras J, Gardovskis J, Vaasna T, Kupcs U, Pupelis G, Dukart G, Dartois N, Jouve S, Cooper A; 305 Study Group. Overview of tigecycline efficacy and safety in the treatment of complicated skin and skin structure infections - a European perspective. J Chemother. 2008 Oct;20 Suppl 1:20-7. doi: 10.1179/joc.2008.20.Supplement-1.20. PMID 19036671